CLINICAL TRIAL: NCT03751878
Title: Evaluating the Impact of Assessing During Peer Review the CONSORT Checklist Submitted by Authors: a Randomised Controlled Trial
Brief Title: Evaluating the Impact of Assessing During Peer Review the CONSORT Checklist Submitted by Authors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Politècnica de Catalunya (Other)
Collaborators: University of Liverpool (Other); The BMJ (Other)
Responsible Party: Principal Investigator, David Blanco, Principal Investigator, Universitat Politècnica de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC 02
Record Dates: First submitted 2018-11-21; First posted 2018-11-23 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Peer Review, Publishing; Completeness of Reporting
Keywords: Reporting guidelines; CONSORT; Adherence; Completeness of reporting; Quality of reporting; Peer review

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Evaluation of reporting inconsistencies between the CONSORT checklist and the information reported in the manuscript. Feedback is provided to authors.
  Interventions: Behavioral: Evaluation of reporting inconsistencies
- Control arm (Other): Standard peer review process.
  Interventions: Behavioral: Standard Peer Review.

INTERVENTIONS:
Behavioral: Evaluation of reporting inconsistencies — 1. The completed CONSORT checklist submitted by authors of manuscripts randomised to the intervention group will be assessed by the lead investigator (DB) as to whether it is consistent with the information that was actually reported in the manuscript. This evaluation will be focused on 8 core CONSORT items.
  2. DB will produce a standardised report containing precise requests for authors in order to improve the completeness of reporting of the items where reporting inconsistencies were found. This report will consist of a brief introduction followed by a point by point description of the inconsistencies found together with precise requests related to the information missing and examples extracted from CONSORT. DB will upload this report to the submission on the managing system of the journal (Scholar One) to make it accessible to the handling editor of the manuscript.
  3. This editor will include the report in the letter to authors alongside the standard peer review reports.
  Arms: Intervention arm
Behavioral: Standard Peer Review. — Manuscripts will undergo the usual peer review process.
  Arms: Control arm

SUMMARY:
Randomised trials are considered the gold standard in medical research. The CONSORT (Consolidated Standards of Reporting Trials) Statement aims to improve the quality of reporting of randomised trials. Without transparent reporting, readers cannot judge the reliability and validity of trial findings, and therefore these findings cannot inform clinical practice. Different stakeholders, including biomedical journals, have taken different actions to try to improve author adherence to CONSORT. The most popular action among biomedical journals is to instruct authors to submit a completed RG checklist with page numbers indicating where the CONSORT items are addressed when they submit their manuscript. However, this measure alone has been proven not to be effective. In this study, the investigators intend to evaluate in a real editorial context whether assessing during peer review the consistency between the submitted CONSORT checklist and the information reported in the manuscripts of randomised trials, as well as to provide feedback to authors on the inconsistencies found, improves the completeness of reporting of published trials.

DETAILED DESCRIPTION:
Randomised trials are considered the gold standard in medical research. The CONSORT (Consolidated Standards of Reporting Trials) Statement aims to improve the quality of reporting of randomised trials. Without transparent reporting, readers cannot judge the reliability and validity of trial findings, and therefore these findings cannot inform clinical practice.

In recent years, different stakeholders have acted to boost the completeness of reporting of the published randomised trials, and therefore their transparency and reproducibility. In a recently completed scoping review, the investigators identified and classified 31 interventions to improve adherence to reporting guidelines. This review revealed that it is primarily journals that have taken most efforts to improve the completeness of reporting of randomised trials - although most of their actions have been shown not to have the desired effect.

One of the most popular strategies used by journals to improve adherence to CONSORT requires authors to submit a populated checklist together with their manuscript indicating page numbers corresponding to each item. However, journals usually lack further actions throughout the editorial process to ensure that the corresponding information to each item is reported in the randomised trial manuscript. This has been hypothesized to be one of the reasons why this editorial strategy has not achieved optimal results.

In an effort to take full advantage of requiring the submission of populated checklists, the investigators intend to evaluate in a real editorial context whether assessing during peer review the consistency between the submitted CONSORT checklist and the information reported in the manuscripts of randomised trials, as well as to provide feedback to authors on the inconsistencies found, improves the completeness of reporting of published trials.

ELIGIBILITY:
Inclusion Criteria:

Manuscripts will be eligible if:

* They have been submitted to BMJ Open,
* They are original research submissions reporting the results of a randomised trial, and
* They have passed the first editorial filters and have been subsequently sent out for peer review.
* Authors of these manuscripts have provided a completed CONSORT checklist.

According to the official CONSORT extensions, the investigators will also consider other study designs (cluster, non-inferiority and equivalence, pragmatic, N-of-1 trials, Pilot and feasibility, and within person trials), and different intervention types (Herbal, non-pharmacologic, acupuncture and Chinese herbal medicine formulas) in all areas of clinical specialty.

Exclusion Criteria:

* Protocols of randomised trials
* Secondary trial analysis studies

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2019-04-13 (Actual); Study Completion 2019-04-13 (Actual)

PRIMARY OUTCOMES:
Overall completeness of reporting | Following manuscript revision (usually 2-3 months)
  Proportion of adequately reported CONSORT items in the first revised manuscript

SECONDARY OUTCOMES:
Completeness of reporting for each item | Following manuscript revision (usually 2-3 months)
  Proportion of manuscripts where each CONSORT item is adequately reported
Time to perform the evaluation | Following the evaluation of reporting inconsistencies (1 week)
  Time to perform the evaluation of reporting inconsistencies by the lead investigator (DB)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Schroter, Study Chair — The BMJ, London; Adrian Aldcroft, Study Chair — The BMJ, London; David Moher, Study Chair — Ottawa Hospital Research Institute, Ottawa; Isabelle Boutron, Study Chair — Paris Descartes University, Paris; Jamie J Kirkham, Study Chair — University of Liverpool, Liverpool; Erik Cobo, Study Chair — Universitat Politècnica de Catalunya, Barcelona
Locations (1):
- BMJ Open, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The content of the interventional peer review reports will appear as part of the review history of the manuscripts. However, in order to protect confidentiality, no dataset including individual manuscript data or outcome data identifying the performance of individual participants will be released. When the study is finished, DB will assign a study number to each paper and store that code with the manuscript ID, password protect it, and store it (File 1) in the BMJ Google Drive folder for the study. In this file, we will also include all identifying variables (Submission date, Trial registration number, Title, Latest editorial decision, applicable CONSORT extensions). For the file containing the peer review reports and the study outcomes (File 2), DB will strip all identifying variables other than the study code and store that file separate from File 1. DB will stick all study files in one folder, compress this folder using WinZip, password protect it, and store it in the same folder.

REFERENCES:
- [Derived] Blanco D, Schroter S, Aldcroft A, Moher D, Boutron I, Kirkham JJ, Cobo E. Effect of an editorial intervention to improve the completeness of reporting of randomised trials: a randomised controlled trial. BMJ Open. 2020 May 18;10(5):e036799. doi: 10.1136/bmjopen-2020-036799. PMID 32430454

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT03751878/Prot_SAP_003.pdf